CLINICAL TRIAL: NCT06637111
Title: Ultrasound Guidance of Office Hysteroscopy in Patients With History of Failure of Office Hysteroscopy Due to Cervical Stenosis.A Randomized Controlled Study
Brief Title: Ultrasound Guidance of Office Hysteroscopy in Patients With History of Failure of Office Hysteroscopy Due to Cervical Stenosis.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Collaborators: Bedaya Hospital (Other)
Responsible Party: Principal Investigator, Usama M Fouda, Prof,, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Ultrasonography/hysteroscopy
Record Dates: First submitted 2024-10-09; First posted 2024-10-15 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Hysteroscopy
Keywords: Hysteroscopy; Ultrasound; Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ultrasound guided office hysteroscopy group (Active Comparator): All the procedures will be performed using the vaginoscopic technique. A rigid 2.9-mm hysteroscope with a 30° lens and a 5-mm outer sheath (Karl Storz GmbH, Tuttlingen, Germany) will be used in all procedures.
  A 5 Fr grasper and 5 Fr scissors will be used to widen the stenotic internal or external ostia.
  Transabdominal ultrasound will be used to guide the access of the hysteroscope to the uterine cavity
  Interventions: Procedure: Ultrasound guided office hysteroscopy group
- Conventional office hysteroscopy group (Active Comparator): All the procedures will be performed using the vaginoscopic technique. A rigid 2.9-mm hysteroscope with a 30° lens and a 5-mm outer sheath (Karl Storz GmbH, Tuttlingen, Germany) will be used in all procedures.
  A 5 Fr grasper and 5 Fr scissors will be used to widen the stenotic internal or external ostia.
  Interventions: Procedure: Conventional office hysteroscopy group

INTERVENTIONS:
Procedure: Ultrasound guided office hysteroscopy group — One hour before office hysteroscopy, 100 mg of diclofenac potassium will be administered per orem. The patients will be asked to drink about one liter of water and to avoid urination before the procedure Moreover, a few minutes prior to the office hysteroscopy, 3 ml of 5% lidocaine and prilocaine topical cream will be introduced into the endocervical canal.
  All procedures will be performed using the vaginoscopic technique. A rigid 2.9-mm hysteroscope with a 30° lens and a 5-mm outer sheath (Karl Storz GmbH, Tuttlingen, Germany) will be used in all procedures.
  A 5 Fr grasper and 5 Fr scissors will be used to widen the stenotic internal or external ostia.
  Transabdominal ultrasound will be used to guide the access of the hysteroscope to the uterine cavity
  Arms: Ultrasound guided office hysteroscopy group
Procedure: Conventional office hysteroscopy group — One hour before office hysteroscopy, 100 mg of diclofenac potassium will be administered per orem . The patients will be asked to drink about one liter of water and to avoid urination before the procedure Moreover, a few minutes prior to the office hysteroscopy, 3 ml of 5% lidocaine and prilocaine topical cream will be introduced into the endocervical canal.
  All the procedures will be performed using the vaginoscopic technique. A rigid 2.9-mm hysteroscope with a 30° lens and a 5-mm outer sheath (Karl Storz GmbH, Tuttlingen, Germany) will be used in all procedures.
  A 5 Fr grasper and 5 Fr scissors will be used to widen the stenotic internal or external ostia.
  Arms: Conventional office hysteroscopy group

SUMMARY:
The study is conducted to assess whether ultrasound guidance can facilitate the access of the office hysteroscope into the uterine cavity of patients with previous failure of office hysteroscopy due to cervical stenosis.

ELIGIBILITY:
Inclusion Criteria:

* Patients with history of failure of office hysteroscopy

Exclusion Criteria:

* Pelvic inflammatory disease
* Severe vaginal bleeding
* Pregnancy
* Allergy to lidocaine, prilocaine or diclofenac potassium

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Estimated)
Dates: Start 2024-10-30 (Actual); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
Success of office hysteroscopy [ ability to gain access of the hysteroscope into uterine cavity] | Immediately after the procedure
  Percentage of successfully performed office hysteroscopy [ = number of successful office hysteroscopies /total number of office hysteroscopies]

SECONDARY OUTCOMES:
Intensity of pain | Immediately after the procedure
  Measured using 100 mm visual analogue scale ( 0 = no pain and 100 = worst possible pain)

CONTACTS AND LOCATIONS:
Overall Officials: Usama M Fouda, Principal Investigator — Cairo University
Locations (2):
- Egypt (2):
  - Faculty of medicine, Cairo university, Cairo
  - Obstetrics &Gynecology Department , Faculty of medicine ,Cairo university, Cairo

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kresowik JD, Syrop CH, Van Voorhis BJ, Ryan GL. Ultrasound is the optimal choice for guidance in difficult hysteroscopy. Ultrasound Obstet Gynecol. 2012 Jun;39(6):715-8. doi: 10.1002/uog.11072. PMID 22173892